CLINICAL TRIAL: NCT06821334
Title: A Randomized, Double-Blind, Placebo-Controlled Single Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics of MK-6194 in Healthy Chinese Participants
Brief Title: A Single Dose Study of MK-6194 in Healthy Chinese Participants (MK-6194-014)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 6194-014; MK-6194-014 (Other: MSD)
Record Dates: First submitted 2025-02-10; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Panel A (Experimental): Participants receive single dose subcutaneous (SC) injection of MK-6194 (Dose 1) or Placebo.
  Interventions: Biological: MK-6194; Biological: Placebo
- Panel B (Experimental): Participants receive single dose subcutaneous (SC) injection of MK-6194 (Dose 2) or Placebo.
  Interventions: Biological: MK-6194; Biological: Placebo
- Panel C (Experimental): Participants receive single dose subcutaneous (SC) injection of MK-6194 (Dose 3) or Placebo.
  Interventions: Biological: MK-6194; Biological: Placebo

INTERVENTIONS:
Biological: MK-6194 — Subcutaneous Administration
Biological: Placebo — Subcutaneous administration

SUMMARY:
The goal of this study is to learn how safe MK-6194 is in healthy Chinese adults and how well people tolerate it.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Is in good health
* Has body mass index (BMI) within 18.0 to 28.0 kg/m^2 (inclusive) and weight ≥50 kg

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* History of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Has a history of opportunistic infection, Human immunodeficiency virus (HIV), hepatitis B, hepatitis C, tuberculosis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2024-04-23 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-08-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to 42 days post dose
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Due to an AE | Up to 42 days post dose
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be reported.

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Last Measurable Concentration (AUC0-Last) of MK-6194 | Up to 42 days post dose
  Blood samples will be collected at specified intervals to determine the AUC0-last of MK-6194.
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of MK-6194 | Up to 42 days post dose
  Blood samples will be collected at specified intervals to determine the AUC0-inf of MK-6194.
Maximum Serum Concentration (Cmax) of MK-6194 | Up to 42 days post dose
  Blood samples will be collected at specified intervals to determine the Cmax of MK-6194.
Time to Maximum Serum Concentration (Tmax) of MK-6194 | Up to 42 days post dose
  Blood samples will be collected at specified intervals to determine the Tmax of MK-6194.
Apparent Terminal Half-life (t1/2) of MK-6194 | Up to 42 days post dose
  Blood samples will be collected at specified intervals to determine the t1/2 of MK-6194.
Apparent Clearance (CL/F) of MK-6194 | Up to 42 days post dose
  Blood samples will be collected at specified intervals to determine the CL/F of MK-6194.
Apparent Volume of Distribution during terminal phase (Vz/F) of MK-6194 | Up to 42 days post dose
  Blood samples will be collected at specified intervals to determine the Vz/F of MK-6194.
Incidence of Antidrug Antibodies (ADA) to MK-6194 | Up to 42 days post dose
  Blood samples will be collected at specified intervals to determine the ADA response to MK-6194.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Peking University Third Hospital (Site 0001), Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com